CLINICAL TRIAL: NCT04981548
Title: Ultrasonography of Optic Nerve Sheath Diameter for Noninvasive Detection of Raised Intracranial Pressure: a Chinese Multicenter Study
Brief Title: Ultrasonography of Optic Nerve Sheath Diameter for Noninvasive Detection of Raised Intracranial Pressure: ORIENT Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, LIJUAN WANG, associate professor, The First Hospital of Jilin University
Other Study IDs: 21K081-001
Record Dates: First submitted 2021-07-26; First posted 2021-07-29 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Ultrasonography
Keywords: optic nerve sheath diameter; intracranial pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- raised intracranial pressure: more than 200 mmH2O
  Interventions: Other: no intervention
- the normal intracranial pressure group: more than 80 mmH2O and no more than 200 mmH2O
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study aims to adopt a multi-center large sample size study to define (1) the normal range of Chinese ONSD; (2) ONSD diagnosis for patients with high intracranial pressure; (3) to analyze the correlation between ONSD and intracranial pressure.

DETAILED DESCRIPTION:
The ONSD, transcranial Doppler parameters and baseline data of the normal intracranial pressure group and the enhanced intracranial pressure group (more than 200 mmH2O) .

ELIGIBILITY:
Inclusion Criteria:

1. People requiring lumbar puncture testing due to brain trauma, intracranial infection, intracranial vascular disease, intracranial tumors, peripheral neuropathy for the raised intracranial pressure group.
2. Healthy people for the normal intracranial pressure group.

Exclusion Criteria:

1. eye diseases, such as eye trauma, eye tumors, optic neuritis, and glaucoma
2. People with poor temporal window penetration.
3. Patients who refuse to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with suspected high intracranial pressure requiring lumbar puncture to measure spinal fluid pressure.
  The normal population is healthy volunteers with matching gender and age, requiring previous physical fitness, has no history of eye diseases, such as eye trauma, eye tumors, optic neuritis, and glaucoma.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-11-06 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
The normal range of ONSD in healthy Chinese adults. | 2021.8-2022.8
  We will perform ONSD measurements with normal people by using ultrasound. We aim to establish the range for optic nerve sheath diameter (ONSD) in healthy Chinese adults. And the normal range of ONSD will be measured and reported.
determine the ONSD cut-off point for high intracranial pressure. | 2021.8-2022.8
  We will perform ONSD measurements with patients who was suspected high intracranial pressure rand enquiring lumbar puncture. We will analyze the correlation between ONSD and intracranial pressure. And ONSD cut-off point for evaluating high intracranial pressure will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- the first hospital of Jilin university, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
the study protocal wil be shared with other researchers.
Supporting Information: Study Protocol
Time Frame: the study protocal will become available on December 2022 and for 2 years.

REFERENCES:
- [Background] Wang LJ, Chen LM, Chen Y, Bao LY, Zheng NN, Wang YZ, Xing YQ. Ultrasonography Assessments of Optic Nerve Sheath Diameter as a Noninvasive and Dynamic Method of Detecting Changes in Intracranial Pressure. JAMA Ophthalmol. 2018 Mar 1;136(3):250-256. doi: 10.1001/jamaophthalmol.2017.6560. PMID 29392301